CLINICAL TRIAL: NCT03301441
Title: Sensitivity to Acute Middle Cerebral or Intracranial Carotid Artery Occlusion in MIGrainers - SAMCO-MIG
Brief Title: Sensitivity to Acute Cerebral Ischemia in Migrainers
Acronym: SAMCO-MIG
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9789
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke; Migraine; Migraine With Aura
Keywords: migraine; migraine with aura; migraine without aura; ischemic stroke; Mismatch
MeSH Terms: conditions — Ischemic Stroke; Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migrainers: Patients experiencing an acute brain infarction complicating the occlusion of the internal carotid artery or the first or second segment of the middle cerebral artery. Migraine status determined by the validated French short questionnaire ef-ID Migraine (Classification into migraine without or with aura)
  Interventions: Other: questionnaire ef-ID Migraine
- Non migrainers: Patients experiencing an acute brain infarction complicating the occlusion of the internal carotid artery or the first or second segment of the middle cerebral artery. Migraine status determined by the validated French short questionnaire ef-ID Migraine A short questionnaire validating the absence of migraine
  Interventions: Other: questionnaire ef-ID Migraine

INTERVENTIONS:
Other: questionnaire ef-ID Migraine — All consecutive patients eligible to the study will be included within 7 days of their initial admission, and evaluated with a short questionnaire classifying them as "migrainers" whose status will undergo a detailed validation at 3 months by a migraine expert, and "non-migrainers" whose status will be validated by repeating the short questionnaire at the follow-up visit at 3 months.
  Initial multimodal imaging, done routinely in any stroke patient, will acquire the raw data necessary to calculate the mismatch ratio (MRI DWI/PWI or CT rCBF/CTP). All radiological data will be analyzed centrally after the end of the recruitment, by investigators blinded to the migraine status.

SUMMARY:
Sensitivity to Acute Middle cerebral or intracranial Carotid artery Occlusion in MIGrainers (SMCO-MIG) is a prospective multi-center study to determine if migraine induces a faster infarct growth as assessed by initial multimodal imaging.

DETAILED DESCRIPTION:
Ischemic stroke results from the occlusion of a brain artery by a clot. Early revascularization by thrombolysis and thrombectomy promotes neurological recovery by saving the area of ischemic penumbra. Progression of ischemic stroke is evaluated on multimodal imaging by the "mismatch ratio" between necrotized core and salvageable hypoperfused volumes.

Migraine affects 12% of the population. Although considered as a benign condition, migraine, particularly with aura, is a risk factor for ischemic stroke. Based on pathophysiological hypothesis and the result of one study, which had several limitations, it's suggest that migraine might increase the sensitivity to cerebral ischemia and induce a faster infarct growth.

The main objective of the study is to determine if the mismatch ratio between irreversibly injured and hypoperfused volumes, measured on initial imaging (MRI or CT) during acute ischemia due to occlusion of the middle cerebral artery or the intracranial internal carotid artery, varies according to the migraine status.

A multicentric prospective cohort will be conduct, outcome study. The initial multimodal imaging (MRI or CT) will be acquired routinely using a harmonized protocol in any patient suspected of an acute stroke. All consecutive patients eligible to the study will be included within 7 days of their initial admission, and evaluated with a short questionnaire classifying them as "migrainers" whose status will undergo a detailed validation at 3 months by a migraine expert, and "non-migrainers" whose status will be validated by repeating the short questionnaire at the follow-up visit at 3 months. All radiological data will be analyzed centrally after the end of the recruitment, by investigators blinded to the migraine status.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 75 years old
* Admitted to a stroke unit for an acute ischemic stroke (<12 h)
* Angiography showing M1/M2 or intracranial internal carotid artery occlusion
* MRI or CT acquired <24h from IS onset, using a harmonized protocol enabling calculation of the mismatch

Exclusion Criteria:

* Individual enrolled into another study protocol with a period of exclusion still running at potential inclusion
* Coma, dementia, linguistic problem or aphasia preventing responding to the migraine questionnaire
* Refusal of participation
* Persons under legal protection, guardianship or curatorship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing an anterior circulation brain infarction complicating the occlusion of the internal carotid artery or the first or second segment of the middle cerebral artery and admitted within 12 hours of onset
Sampling Method: Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Mismatch ratio (MRI DWI/PWI or CT rCBF/CTP) | 24 hours
  Raw data acquired on initial multimodal imaging done routinely, using a harmonized protocol in any patient suspected of an acute stroke before the enrollment in the study. The mismatch ratio will be calculated after recruitement completion by investigators blinded to the migraine status.

SECONDARY OUTCOMES:
Proportion of patients with no-mismatch pattern on initial imaging | 24 hours
  ratio DWI/PWI or rCBF/CTP > 0.83
Proportion of patients treated by recanalisation | 24 hours
  thrombolysis and/or thrombectomy
Volume of brain infarction | 24 hours
  Volume of brain infarction 24 hours after thrombolysis and/or thrombectomy
TICI score | 24 hours
  Quality of revascularization after thrombolysis and/or thrombectomy
Modified Rankin Score | 3 months
  Good functional outcome will be defined by a Modified Rankin Scale of 0-2, 3 months after stroke onset
Modified Rankin Score in patients treated by thrombolysis and/or thrombectomy | 3 months
  Good functional outcome will be defined by a Modified Rankin Scale of 0-2, 3 months after stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Anne DUCROS, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier - Neurology Departement, Montpellier, France